CLINICAL TRIAL: NCT03295292
Title: Pilot Clinical Trial to Assess the Safety of Limbus-derived Corneal Stem Cells in Prevention of Corneal Haze After Photo Therapeutic/Refractive Keratectomy (PTK/ PRK) and Collagen Cross Linking (CXL)
Brief Title: Limbus-derived Stem Cells for Prevention of Postoperative Corneal Haze
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, Vivek Singh, Prinicipal Investigator, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEC 07-17-068
Record Dates: First submitted 2017-08-19; First posted 2017-09-27 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Corneal Scars and Opacities
Keywords: Phototherapeutic Keratectomy (PTK); photorefractive Keratectomy (PRK); Collagen Cross-linking (CXL); Stem Cell Therapy
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Surgery with Vehicle (Sham Comparator): After the standard surgical procedure (PRK/PTK or CXL), patients will receive 50uL Fibrin Sealant (sham) without cells.
  Interventions: Other: Vehicle
- Standard Surgery with Stem Cells (Experimental): After the standard surgical procedure (PRK/PTK or CXL), patients will receive 50uL of a mixture of limbus derived corneal epithelial cells and limbus derived corneal stromal cells in a ratio of 2:1, at a concentration of 50000 cells/uL diluted in the thrombin component of Fibrin Sealant (TISEEL, Baxter).
  Interventions: Biological: Stem cells; Other: Vehicle

INTERVENTIONS:
Biological: Stem cells — Mixture of limbus derived corneal epithelial cells and limbus derived corneal stromal cells in a ratio of 2:1, at a concentration of 50000 cells/uL diluted in fibrin sealant
  Arms: Standard Surgery with Stem Cells
Other: Vehicle — 50uL of commercially available fibrin sealant (Baxter, TISEEL)

SUMMARY:
This is a investigator-initiated pilot clinical trial to ascertain the safety and efficacy of application of ex-vivo cultivated limbal stem cells in human eyes for treating Corneal Haze after Photo-Therapeutic/Refractive Keratectomy (PTK/ PRK) and Collagen Cross Linking (CXL). Instead of using adjunctive medical therapy like application of MMC (Mitomycin), a technique of cell delivery with fibrin sealant can be used. These cells are harvested from therapeutically accepted and serologically tested cadaveric corneas. The isolated limbal epithelial and mesenchymal or stromal cell suspension will then be cultured in CGMP laboratories and be tested for sterlity. These cells have also been shown to be effective in treating haze in laser refractive surgery in an animal model. Our initial experience of using these cells in a previous clinical trial showed that they were effective in preventing corneal haze in patients with burns and ulcers.

DETAILED DESCRIPTION:
In this pilot clinical trial, patients undergoing Photo Therapeutic/Refractive Keratectomy (PTK/ PRK) and Collagen Cross Linking (CXL), will be given human Limbus-derived Corneal Stem cells to assess the safety of these cells. Cells will be cultivated in a cGMP laboratory using standardized culture technique; from the limbal rims of cadaveric corneoscleral donor tissues that are therapeutically accepted and serologically tested. Briefly the limbal tissue will be cut up into small pieces and digested overnight using an enzyme (Collagenase L). The cells obtained from the digest will be cultured on a petri-dish using 2% serum and growth factors. A mixture of limbal epithelial cells and limbal stromal cells obtained from these cultures will be used in surgical procedures in a ratio of 2:1, after all the sterility checks. Mixed suspension of the limbal epithelial and the stromal cells at a concentration of 50000 cells/uL diluted in the thrombin component of fibrin sealant (TISEEL, Baxter) will be applied. The primary outcome measure is safety of this treatment and the secondary outcome measure is their efficacy that will be assessed at 1 month time points by (1) Clinical photography using a standard method where multiple blinded observers will grade the clinically apparent change in haze and (2) Objective quantification of the amount of light scattering using densitometry analysis function in Oculus Pentacam (OCULUS Optikgeräte GmbH).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between20 to 40 years of age
* Meeting standard selection criteria for bilateral PTK/PRK or CXL
* No systemic diseases
* Eligible to give informed consent
* No other ocular co-existing pathologies

Exclusion Criteria:

* Undergoing surgery in only one eye
* Grossly asymmetric pathology
* Refusal to give informed consent
* Not agreeable or uncooperative for corneal imaging
* Unlikely to come for follow-up for 1 month
* International and out-station patients

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Maintenance of pre-operative best-spectacle corrected visual acuity | 1 month

SECONDARY OUTCOMES:
Efficacy in reducing corneal light scatter using Scheimpflug imaging | 1 month
  Efficacy in reducing corneal light scatter using Scheimpflug imaging at 1 month by:
  Objective quantification of the amount of light scattering using densitometry analysis function in Oculus Pentacam (OCULUS Optikgeräte GmbH).
  • All routine clinical and imaging protocols performed for patients undergoing PTK/PRK and CXL will be diligently followed.

CONTACTS AND LOCATIONS:
Overall Officials: Sayan Basu, MBBS MS, Principal Investigator — LV Prasad Eye Institute; Vivek Singh, MSc PhD, Principal Investigator — LV Prasad Eye Institute; Jagadesh C Reddy, MBBS MD, Principal Investigator — LV Prasad Eye Institute; Pratik Gogri, MBBS MS, Principal Investigator — LV Prasad Eye Institute
Locations (1):
- LV Prasad Eye Institute, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Basu S, Hertsenberg AJ, Funderburgh ML, Burrow MK, Mann MM, Du Y, Lathrop KL, Syed-Picard FN, Adams SM, Birk DE, Funderburgh JL. Human limbal biopsy-derived stromal stem cells prevent corneal scarring. Sci Transl Med. 2014 Dec 10;6(266):266ra172. doi: 10.1126/scitranslmed.3009644. PMID 25504883
- [Result] Basu S, Damala M, Singh V. Limbal Stromal Stem Cell Therapy for Acute and Chronic Superficial Corneal Pathologies: Early Clinical Outcomes of The Funderburgh Technique. Investigative Ophthalmology & Visual Science. 2017 Jun 23;58(8):3371-337